CLINICAL TRIAL: NCT06478901
Title: Precision and RElevance of CardIac ultraSound Using Artificial Intelligence for Left Ventricle Ejection Fraction Assessment in the Elderly. ( PRECISE AI)
Brief Title: Precision of AI-Based Cardiac Ultrasound for LVEF in the Elderly
Acronym: PRECISE AI
Status: Completed | Type: Observational
Sponsor: Hôpital Broca APHP (Other)
Responsible Party: Sponsor
Other Study IDs: PRECIS-AI-2024-01
Record Dates: First submitted 2024-06-10; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure; Heart Failure Systolic; Elderly; Artificial Intelligence
Keywords: Elderly; Left ventricular ejection fraction; Artificial intelligence; Echocardiography
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 129 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiography — Echocardiography assited by Artificial intelligence

SUMMARY:
Heart failure (HF) is common in older adults, especially those over 65. It is a leading cause of hospitalization and has high mortality rates. Diagnosing HF in elderly patients can be challenging due to atypical symptoms and multiple other health issues. Echocardiography, an ultrasound of the heart, is crucial for accurate diagnosis and treatment planning.

One problem in geriatric care is the difficulty of accessing echocardiography due to high demand and limited specialized doctors. Recent advancements show that AI-assisted portable ultrasound devices can reliably measure heart function, producing results comparable to traditional methods.

This study aims to evaluate the accuracy and relevance of AI-assisted echocardiography (AutoEF-AI) in elderly patients. It also assesses whether geriatricians, even without specialized training, can capture quality images for AI analysis.

In simple terms, this study investigates if portable ultrasound devices with AI can provide precise heart function diagnostics, making it easier for older adults with heart failure to get the care they need, even without specialists.

DETAILED DESCRIPTION:
Heart failure (HF) is a major chronic illness, particularly common in older adults. With advances in healthcare and an aging population, HF is increasingly affecting people over 65 years old. In fact, 80% of HF patients are over 65. HF is associated with high mortality rates and is the leading cause of hospitalization after age 80, and even after age 65 in some countries like France.

In older adults, HF symptoms are often atypical due to multiple other health conditions, increased frailty, and associated geriatric syndromes, making diagnosis difficult. In this context, echocardiography (an ultrasound of the heart) is essential for accurately diagnosing HF.

Evaluating the left ventricular ejection fraction (LVEF) through echocardiography is a fundamental step in diagnosing HF and deciding on treatment strategies. This evaluation helps refine the HF diagnosis, propose appropriate treatments, and monitor changes in heart function over time.

One major challenge in geriatric units and nursing homes (EHPADs) is the difficulty in accessing echocardiography due to growing demand and a limited number of specialized doctors.

Recent studies have shown that automated LVEF measurements assisted by artificial intelligence (AI) using portable ultrasound devices are reliable and produce results comparable to traditional methods. This AI-assisted automatic LVEF calculation (AutoEF-AI) could be a major advantage in geriatric departments, providing a credible alternative to conventional echocardiography for evaluating LVEF in HF patients.

The main goal of this study was to evaluate the relevance and accuracy of AutoEF-AI echocardiography in elderly patients. The secondary goal was to assess whether geriatricians without specialized training in echocardiography could capture images of sufficient quality to be analyzed by automatic LVEF algorithms with acceptable accuracy.

In simple terms, this study aims to determine if using portable ultrasound devices, assisted by artificial intelligence, can provide diagnostics as precise as traditional methods. This could make evaluating heart function more accessible and effective for older adults with heart failure, even when specialists are not available.

ELIGIBILITY:
Inclusion Criteria:

* At least 75 years and a clinical presentation of acute heart failure consistent with the criteria of the European Society of Cardiology guidelines

Exclusion Criteria:

* unstable patient

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 75 years or more and a clinical presentation of acute heart failure
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2023-01-14 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
evaluate the relevance and accuracy of echocardiography assisted by Artificial intelligence in elderly patients | From enrollment to the end 48 hours
  The correlation between LVEF measurements from standard echocardiography and AutoEF-AI echocardiography was assessed using the intraclass correlation coefficient (ICC) and Bland-Altman analysis. Weighted Kappa coefficient was calculated to determine agreement between measurements in classifying patients into different categories based on LVEF

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Broca, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.aphp.fr/contenu/hopital-broca-2

REFERENCES:
- [Result] Chaudhry SI, Wang Y, Gill TM, Krumholz HM. Geriatric conditions and subsequent mortality in older patients with heart failure. J Am Coll Cardiol. 2010 Jan 26;55(4):309-16. doi: 10.1016/j.jacc.2009.07.066. PMID 20117435